CLINICAL TRIAL: NCT05500716
Title: The Effect of Application of Vagus Nerve Stimulation on the Treatment Efficiency in Temporomandibular Joint Dysfunction Caused by Myofascial Pain Syndrome
Brief Title: The Effect of Vagus Nerve Stimulation on Temporomandibular Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alper Percin (Other)
Responsible Party: Sponsor-Investigator, Alper Percin, Principle İnvestigator, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDYAP0001
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome; Autonomic Nervous System Imbalance
Keywords: Vagus Nerve Stimulation; Neuromodulation
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Intervention Model Description: All groups will be involved physical therapy and both groups will have traditional rehabilitation program for TMD. Only the group 1 will also have auricular non-invasive vagus nerve stimulation.
Who Masked: Participant
Masking Description: Participants will not be informed about which treatment was given in the other group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auricular Non-Invasive Vagus Nerve Stimulation+Traditional Rehabilitation Program (Experimental): * Auricular Non-Invasive Vagus Nerve Stimulation
  * Deep Friction Massage
  * Myofascial Trigger Point Compression Therapy
  * Temporomandibular Joint Mobilization
  * Rocabado Exercises
  * Muscle-Energy Techniques
  Interventions: Other: Auricular Non-Invazive Vagus Nerve Stimulation + Traditional Rehabilitation Program for TMD
- Traditional Rehabilitation Program (Active Comparator): * Deep Friction Massage
  * Myofascial Trigger Point Compression Therapy
  * Temporomandibular Joint Mobilization
  * Rocabado Exercises
  * Muscle-Energy Techniques
  Interventions: Other: Traditional Rehabilitation Program

INTERVENTIONS:
Other: Auricular Non-Invazive Vagus Nerve Stimulation + Traditional Rehabilitation Program for TMD — In this application, vagus nerve stimulation is applied to the patients in addition to the traditional rehabilitation program. In our research, vagal nerve stimulation will be applied with the "Vagustim" Device and all applications will be applied at a frequency of 10 Hz, a pulse amplitude of 300 microseconds and for 20 minutes.
  Arms: Auricular Non-Invasive Vagus Nerve Stimulation+Traditional Rehabilitation Program
Other: Traditional Rehabilitation Program — This intervention includes: Deep Friction Massage, Myofascial Trigger Point Compression Therapy, Temporomandibular Joint Mobilization, Rocabado Exercises, Muscle-Energy Techniques.
  Arms: Traditional Rehabilitation Program

SUMMARY:
Temporomandibular joint dysfunction (TMD) is a broad clinical picture involving the TMJ and its disc, masticatory musculature, ligament tissue, and autonomic nervous system (ANS). TMD symptoms include decrease or excessive increase in joint range of motion (ROM), clicking sound or crepitation in the joint, pain around the joint or muscle group, chewing and swallowing problems. Pain caused by MPS, trigger point, fatigue, limitation of ROM, and ANS dysfunction cause TMD. With the inclusion of habits such as clenching and bruxism, pain, spasm and disability develop in the chewing muscles. Exposure to repeated trauma and excessive use of chewing muscles may cause the formation of tight bands and trigger points, which are characterized by MPS. When the relationship between TMD and ANS was examined, it was observed that increased sympathetic activity and decreased parasympathetic activity were effective in the severity of TMD symptoms. Auricular vagus nerve stimulation is a peripheral, non-pharmacological and non-invasive neuromodulation technique that modifies signal processing in the CNS, activates reflex circuits, exploits brain plasticity for different therapeutic purposes, thereby affecting very different areas of the brain. Non-invasive or transcutaneous Vagus Nerve Stimulation delivery systems provide stimulation in the auricular branch of the vagus nerve in the outer ear, thus eliminating the need for surgical implantation. The aim of our study is to reveal the extent to which Auricular Vagus Nerve Stimulation, applied in addition to the conventional rehabilitation program, affects the results of the treatment by stimulating the parasympathetic nervous system in patients with Temporomandibular Joint Dysfunction caused by Myofascial Pain Syndrome.

DETAILED DESCRIPTION:
The temporomandibular joint (TMJ) is a ginglymoarthrodial joint, a term derived from ginglymus, meaning a hinge joint that allows only forward and backward movement in one plane, and arthrodia, a joint that allows gliding motion, and right and left TMJ are similar to knee articulation. It forms the ellipsoid variety of bicondylar articulation and synovial joints. TMJ movements are defined as elevation, depression, protrusion, retrusion, and lateralization. Primary muscle groups that reveal these joint movements m. masseter, m. temporalis, medial and lateral pterygoid, suprahyoid (digastricus, mylohyoid, geniohyoid, stylohyoid) and infrahyoid (thyrohyoid, sternohyoid, sternothyroid, omohyoid). The TMJ ligament complex consists of superficial and deep collateral ligament, sphenomandibular ligament and stylomandibular ligament. While the sensory nerves of the TMJ branch from the Trigeminal (V. Cranial nerve) nerve, they receive sympathetic innervation from the cervical ganglion (C8-T3). Temporomandibular joint dysfunction (TMD) is a broad clinical picture involving the TMJ and its disc, masticatory musculature, ligament tissue, and autonomic nervous system (ANS). TMD symptoms include decrease or excessive increase in joint range of motion (ROM), clicking sound or crepitation in the joint, pain around the joint or muscle group, chewing and swallowing problems. TMD is considered in two groups as articular and non-articular disorders: articular disorders express the dislocation of the disc with and without reduction, while non-articular disorders express the problems caused by myofascial pain syndrome (MPS). Pain caused by MPS, trigger point, fatigue, limitation of ROM, and ANS dysfunction cause TMD. With the inclusion of habits such as clenching and bruxism, pain, spasm and disability develop in the chewing muscles. Exposure to repetitive trauma and overuse of chewing muscles may cause the formation of tight bands and trigger points, which are characterized by MPS.

ANS is part of the peripheral nervous system (PSS), which regulates involuntary physiological processes such as heart rate, blood pressure, respiration, and digestion, and is anatomically composed of 3 parts: the sympathetic, parasympathetic, and enteric nervous systems. The sympathetic nervous system (SNS) and parasympathetic nervous system (PNS) contain afferent and efferent pathways that provide sensory and motor stimulation, and these pathways consist of preganglionic neurons in the central nervous system (CNS) and postganglionic neurons in the periphery. The SNS enables the body to handle stressors through the "fight or flight" response, and this reaction primarily regulates the blood vessels. The vessels are tonically innervated and in most cases an increase in sympathetic signals leads to vasoconstriction. SNS activation increases heart rate and contraction force. The PNS exits the SNS via cranial nerves III, VII, IX, and X, as well as via S2-4 nerve roots. The vagus nerve (Cranial Nerve X), together with the sacral parasympathetic fibers, provides parasympathetic input to most of the thoracic and abdominal organs and has four cell bodies: Dorsal nucleus (parasympathetic stimulation of viscera), Nucleus ambiguous (preganglionic neurons innervating the heart), Nucleus solitarius (taste sense) and Trigeminal nucleus (outer ear circumference receives touch, pain and temperature information). The vagus nerve is responsible for the "resting and digesting" processes. By providing cardiac relaxation, the vagus nerve reduces contraction in the atria and ventricles and decreases the conduction velocity through the atrioventricular node. The vagus nerve also has a significant effect on the respiratory cycle, and its activity increases during expiration, constricting and stiffening the airways to prevent lung collapse.

When the relationship between TMD and ANS was examined, it was observed that increased sympathetic activity and decreased parasympathetic activity were effective in the severity of TMD symptoms. It has been shown that TMD patients may show changes in the sympathoadrenal and inflammatory cytokine function resulting from their response to the stressor, and that the increase in the sympathetic activity of these patients in the long term may cause decreased interleukin-6 (IL-6) and norepinephrine response. It is thought that IL-6 may be an important factor related to the increased morbidity and mortality in people with chronic stress and may play a pathogenic role in the course of stress-reactive chronic diseases. Another mechanism thought to cause TMD is that the junctional region between the trigeminal subnucleus caudalis (Vc) and the upper cervical spinal cord, called the Vc/C1-2 region, is the primary site for synaptic integration of sensory input from TMJ nociceptors, and Vc/C1- It is known that estrogen hormone is effective on the processing of nociceptive stimulus by neurons in region 2. Especially in the post-menopausal period, the decrease in the level of estrogen in the blood causes an increase in sympathetic activity and causes pain and disability around the TMJ. Another method of evaluating the relationship between TMD and ANS is the measurement of heart rate variability (HRV). In a study, it was observed that HRV, which is a marker of ANS dysfunction, decreased in patients with myofascial temporomandibular disorder (TMD) compared to healthy individuals.

Auricular vagus nerve stimulation is a peripheral, non-pharmacological and non-invasive neuromodulation technique that modifies signal processing in the CNS, activates reflex circuits, exploits brain plasticity for different therapeutic purposes, thereby affecting very different areas of the brain. Modulation of the afferent vagus nerve affects numerous physiological processes and bodily states associated with the transfer of information between the brain and the body. These include disease mitigating effects and sustainable therapeutic practices ranging from chronic pain diseases, neurodegenerative and metabolic disorders to inflammatory and cardiovascular diseases. Non-invasive or transcutaneous Vagus Nerve Stimulation delivery systems provide stimulation in the auricular branch of the vagus nerve in the outer ear, thus eliminating the need for surgical implantation. One of the non-invasive Vagus Nerve Stimulators in use today, NEMOS®, stimulates the outer ear turbinate and is European Conformity (CE) marked for the European Union for the management of epilepsy. The electrode is connected to a stimulation box and the stimulation intensity can be adjusted by the patient, caregiver, or treating healthcare professional. During use, it is increased in 0.1 milliamperes(mA) steps until the detection threshold of electrical stimulation is reached; the stimulation frequency was defined as 25 Hz. Another non-invasive Vagus Nerve Stimulator gammaCore® is used for transcutaneous stimulation of the cervical branch of the vagus nerve and is FDA approved for the treatment of episodic cluster headache. The device generates a wave in the form of a pulse. It creates impulses with a 1 ms transition time of an electrical current with a frequency of 25 Hz. The recommended stimulation time is 2 minutes and can be applied up to 12 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Compliant with temporomandibular disorders research/diagnosis criteria,
* Diagnosed with Myofascial Pain Syndrome,
* 18 years and over,
* Female patients who volunteered to participate in the study and filled in the informed consent form will be included in the study.

Exclusion Criteria:

* History of TMJ disc dislocation,
* History of acute trauma in and around the TMJ,
* Having a history of surgical/invasive procedures on the TMJ,
* Having a neurological or psychiatric diagnosis,
* Being pregnant,
* Presence of infection or tumoral structure within intraoral structures
* Having a history of tooth loss, use of prosthetic teeth,
* Having a history of surgical procedures in the cervical region,
* Previous treatment related to TMD,
* be under the age of 18,
* Participants will be excluded from the study if they are in the post-menopausal stage.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | Measurements will be completed between beginning-4 weeks-8 weeks-12 weeks
  Heart rate variability (HRV) is a popular, non-invasive, physiological assessment tool among clinicians for monitoring ANS activity. Studies have shown how clinicians can examine the magnitude of autonomic modulation by examining the variability between resting heart rate (HR) and beat-beat (RR) intervals in response to training stress or psychological stress.Heart rate variability will be measured with the polar h10 device.

SECONDARY OUTCOMES:
Pain and Trigger Points | Measurements will be completed between beginning-4 weeks-8 weeks-12 weeks
  It is applied to Temporalis and masseter muscles, posterior mandible region and submandibular region in the evaluation of trigger point in temporomandibular region muscles. Trigger point assessment in cervical region muscles is applied to sternocleidomastoideus muscle, scalene muscle, upper trapezius, levator scapula, suboccipital region
Range of motion | Measurements will be completed between beginning-4 weeks-8 weeks-12 weeks
  The temporomandibular joint range of motion will be measured. Mandibular depression, mandibular protrusion and mandibular lateral deviation will be included in this measurements.
Perceived Stress scale | Measurements will be completed between beginning-4 weeks-8 weeks-12 weeks
  The Perceived Stress Scale (PSS) is a classic stress assessment tool and scale used to help us understand how different situations affect our emotions and our perceived stress. Questions on this scale ask about your feelings and thoughts in the last month. It consists of 10 items and each item is scored with a number between 0-4. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Neck Disability Index | Measurements will be completed between beginning-4 weeks-8 weeks-12 weeks
  The Neck Disability Index (BDI) was designed to evaluate how neck pain affects activities of daily living. The questionnaire consisting of 10 questions in total, each question is scored in the range of 0-5 points, with no disability (0-4 points), mild disability (5-14 points), moderate disability (15-24 points), severe disability (25-34). is evaluated as completely disabled (35 and above points).

CONTACTS AND LOCATIONS:
Overall Officials: Hande Başat, M.D., Study Director — Bahçeşehir University
Locations (1):
- Bahçeşehir University, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kisilewicz A, Janusiak M, Szafraniec R, Smoter M, Ciszek B, Madeleine P, Fernandez-de-Las-Penas C, Kawczynski A. Changes in Muscle Stiffness of the Trapezius Muscle After Application of Ischemic Compression into Myofascial Trigger Points in Professional Basketball Players. J Hum Kinet. 2018 Oct 15;64:35-45. doi: 10.2478/hukin-2018-0043. eCollection 2018 Sep. PMID 30429897
- [Background] Ishii H, Koga H, Takanishi A, Katsumata A. Development and experimental evaluation of Oral Rehabilitation Robot that provides maxillofacial massage to patients with oral disorders. Int J Robotics Res. 2009;28:May 19. DOI: doi:10,1177/0278364909104295
- [Result] Gillespie BR. Assessment and treatment of TMJ muscles, fascia, ligaments, and associated structures. Cranio. 1990 Jan;8(1):51-4. doi: 10.1080/08869634.1990.11678300. PMID 2098188
- [Result] Ohrbach R, Dworkin SF. Five-year outcomes in TMD: relationship of changes in pain to changes in physical and psychological variables. Pain. 1998 Feb;74(2-3):315-26. doi: 10.1016/s0304-3959(97)00194-2. PMID 9520246
- [Result] Dworkin SF, LeResche L. Research diagnostic criteria for temporomandibular disorders: review, criteria, examinations and specifications, critique. J Craniomandib Disord. 1992 Fall;6(4):301-55. No abstract available. PMID 1298767
- [Result] Travell JG, Simons DG. Myofascial pain and dysfunction: The trigger point manual. Baltimore: Williams and Wilkins; 5-90,1983.
- [Result] Ohrbach R, Michelotti A. The Role of Stress in the Etiology of Oral Parafunction and Myofascial Pain. Oral Maxillofac Surg Clin North Am. 2018 Aug;30(3):369-379. doi: 10.1016/j.coms.2018.04.011. Epub 2018 Jun 1. PMID 29866454
- [Result] Eisenlohr-Moul TA, Crofford LJ, Howard TW, Yepes JF, Carlson CR, de Leeuw R. Parasympathetic reactivity in fibromyalgia and temporomandibular disorder: associations with sleep problems, symptom severity, and functional impairment. J Pain. 2015 Mar;16(3):247-57. doi: 10.1016/j.jpain.2014.12.005. Epub 2014 Dec 24. PMID 25542636
- [Result] Costello NL, Bragdon EE, Light KC, Sigurdsson A, Bunting S, Grewen K, Maixner W. Temporomandibular disorder and optimism: relationships to ischemic pain sensitivity and interleukin-6. Pain. 2002 Nov;100(1-2):99-110. doi: 10.1016/s0304-3959(02)00263-4. PMID 12435463
- [Result] Tashiro A, Bereiter DA. The effects of estrogen on temporomandibular joint pain as influenced by trigeminal caudalis neurons. J Oral Sci. 2020 Mar 28;62(2):150-155. doi: 10.2334/josnusd.19-0405. Epub 2020 Mar 4. PMID 32132330
- [Result] Eze-Nliam CM, Quartana PJ, Quain AM, Smith MT. Nocturnal heart rate variability is lower in temporomandibular disorder patients than in healthy, pain-free individuals. J Orofac Pain. 2011 Summer;25(3):232-9. PMID 21837290
- [Result] Kaniusas E, Kampusch S, Tittgemeyer M, Panetsos F, Gines RF, Papa M, Kiss A, Podesser B, Cassara AM, Tanghe E, Samoudi AM, Tarnaud T, Joseph W, Marozas V, Lukosevicius A, Istuk N, Sarolic A, Lechner S, Klonowski W, Varoneckas G, Szeles JC. Current Directions in the Auricular Vagus Nerve Stimulation I - A Physiological Perspective. Front Neurosci. 2019 Aug 9;13:854. doi: 10.3389/fnins.2019.00854. eCollection 2019. PMID 31447643
- [Result] Ben-Menachem E, Revesz D, Simon BJ, Silberstein S. Surgically implanted and non-invasive vagus nerve stimulation: a review of efficacy, safety and tolerability. Eur J Neurol. 2015 Sep;22(9):1260-8. doi: 10.1111/ene.12629. Epub 2015 Jan 23. PMID 25614179
- [Result] Jeong KH, Kim ME, Kim HK. Temporomandibular disorders and autonomic dysfunction: Exploring the possible link between the two using a questionnaire survey. Cranio. 2023 Sep;41(5):467-477. doi: 10.1080/08869634.2021.1872313. Epub 2021 Jan 11. PMID 33427101
- [Result] Monaco A, Cattaneo R, Mesin L, Ciarrocchi I, Sgolastra F, Pietropaoli D. Dysregulation of the autonomous nervous system in patients with temporomandibular disorder: a pupillometric study. PLoS One. 2012;7(9):e45424. doi: 10.1371/journal.pone.0045424. Epub 2012 Sep 18. PMID 23028999
- [Result] Robinson LJ, Durham J, MacLachlan LL, Newton JL, Autonomic function in chronic fatigue syndrome with and without painful temporomandibular disorder. Pages 205-219 | Received 22 May 2015, Accepted 28 Aug 2015, Published online: 05 Oct 2015. https://doi.org/10.1080/21641846.2015.1091152
- [Result] Gomes NC, Berni-Schwarzenbeck KC, Packer AC, Rdrigues-Bigaton D. Effect of cathodal high-voltage electrical stimulation on pain in women with TMD. Rev Bras Fisioter. 2012 Jan-Feb;16(1):10-5. English, Portuguese. PMID 22441222
- [Result] Blanco-Aguilera A, Blanco-Hungria A, Biedma-Velazquez L, Serrano-Del-Rosal R, Gonzalez-Lopez L, Blanco-Aguilera E, Segura-Saint-Gerons R. Application of an oral health-related quality of life questionnaire in primary care patients with orofacial pain and temporomandibular disorders. Med Oral Patol Oral Cir Bucal. 2014 Mar 1;19(2):e127-35. doi: 10.4317/medoral.19061. PMID 24121906
- [Result] Gil-Martinez A, Paris-Alemany A, Lopez-de-Uralde-Villanueva I, La Touche R. Management of pain in patients with temporomandibular disorder (TMD): challenges and solutions. J Pain Res. 2018 Mar 16;11:571-587. doi: 10.2147/JPR.S127950. eCollection 2018. PMID 29588615
- [Result] Vijila JY. (2016). Effectiveness of Muscle Energy Technique and Rocabado Exercise Versus Therapeutic Jaw Exercises for Temporomandibular Joint Dysfunction (Doctoral dissertation, Nandha College of Physiotherapy, Erode).
- [Derived] Percin A, Basat H, Ozden AV, Yenisehir S. The effect of auricular vagus nerve stimulation in women with temporomandibular joint disorders: a randomized controlled study. Rev Assoc Med Bras (1992). 2025 Jun 2;71(4):e20241739. doi: 10.1590/1806-9282.20241739. eCollection 2025. PMID 40465996